CLINICAL TRIAL: NCT07020364
Title: Feasibility and Safety of a Single Working Element for Bipolar and Laser Enucleation in Prostate Surgery: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Omar, Assistant professor, Menoufia University
Other Study IDs: Enucleation of prostate
Record Dates: First submitted 2024-11-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Prostate; BPH (Benign Prostatic Hyperplasia)
Keywords: laser enucleation; bipolar enucleation; BPH; prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bipolar Enucleation: Bipolar Enucleation Group: The bipolar energy will be used for cutting and coagulation during enucleation.
  Interventions: Device: A single working element for bipolar enucleation
- Laser Enucleation: Laser Enucleation Group: Thulium or Holmium laser will be employed for tissue dissection and hemostasis.
  Interventions: Device: A single working element for laser enucleation

INTERVENTIONS:
Device: A single working element for bipolar enucleation — Device: A single working element compatible with both bipolar and laser modalities.
  The bipolar energy will be used for cutting and coagulation during enucleation.
  Groups: Bipolar Enucleation
Device: A single working element for laser enucleation — Device: A single working element compatible with both bipolar and laser modalities.
  Thulium or Holmium laser will be employed for tissue dissection and hemostasis.
  Groups: Laser Enucleation

SUMMARY:
A prospective feasibility study would be a practical first step, focusing on real-time assessment and ensuring the new working element's integration is safe and effective before broader clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with benign prostatic hyperplasia (BPH) requiring surgical intervention.
* Prostate volume ≥40 cc (as assessed by transrectal ultrasound).
* No prior history of prostate cancer.

Exclusion Criteria:

* Patients with ongoing urinary tract infections.
* Prior prostate surgeries.
* Coagulation disorders or patients on long-term anticoagulation therapy.
* Known urethral strictures or other anatomical abnormalities complicating endoscopic procedures.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study will include male patients aged ≥50 years who are diagnosed with benign prostatic hyperplasia (BPH) , prostate volume ≥40 cc without 4prior history of prostate cancer while patients with ongoing urinary tract infections, prior prostate surgeries, coagulopathy or urethral strictures were excluded.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | the operative time
  Successful completion of enucleation using the single working element. Time taken to switch between bipolar and laser modalities.
Safety | 1 month
  intraoperative complications (bleeding, urethral damage). Postoperative complications (infections, catheterization time, hospital stay).

SECONDARY OUTCOMES:
Efficacy | 1 month
  Operative time. Enucleation efficiency (grams of tissue removed per minute). Postoperative symptom improvement measured using International Prostate Symptom Score (IPSS).
Cost Analysis | the operative time
  Cost of using a single working element vs. standard separate tools for bipolar and laser.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shibīn al Kawm, Menoufia, Egypt